CLINICAL TRIAL: NCT05330364
Title: Clinical Study of Efficacy and Safety of Chidamide Combined With Cladribine Regimen in Refractory/Relapsed Acute Myeloid Leukemia
Brief Title: Study of Chidamide Combined With Cladribine in Refractory/Relapsed Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ge Zheng (Other)
Responsible Party: Sponsor-Investigator, Ge Zheng, Director of Department of Hematology, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDYYGZ202103
Record Dates: First submitted 2022-03-22; First posted 2022-04-15 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Chidamide; Cladribine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Cladribine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide plus Cladribine (Experimental): Chidamide 30mg/d per os (p.o.), twice per week, begins at day 1; Cladribine 5mg/m2/d, intravenous injection (i.v.), days 1-5, once per day; A cycle is during 28 days.
  Interventions: Drug: Chidamide; Drug: Cladribine

INTERVENTIONS:
Drug: Chidamide — Chidamide 30mg/d p.o. begin at day 1, twice per week, during a 28-days cycle.
Drug: Cladribine — Cladribine 5mg/m2/d i.v. d1-5, once per day, during a 28-days cycle.

SUMMARY:
Acute myeloid leukemia (AML) is highly heterogeneous, the efficacy of the individual varies greatly, and the risk of recurrence is high. A large number of newly diagnosed AML patients cannot achieve complete remission (CR) after standard induction chemotherapy. The prognosis of AML patients after relapse is extremely poor, and only a few patients can get remission through salvage treatment.

Chidamide is a histone deacetylase inhibitor (HDACi) independently developed by China. It has been marketed in recent years and the first innovative drug approved by the U.S. Food and Drug Administration for clinical research in the United States. Chidamide can increase the sensitivity of leukemia cells to conventional chemotherapy by inhibiting cell proliferation, inducing apoptosis, and increasing cell cycle arrest. Chidamide and other drugs have different effects in combination, and jointly bear the anti-tumor effect, which provides a theoretical basis for Chidamide in the treatment of acute myeloid leukemia.

Cladribine is a purine nucleoside analog, which has the ability to inhibit DNA synthesis, repair, induce apoptosis, and has anti-leukemia activity for cells in both mitotic and quiescent phases. In the past ten years, many studies have proved that Cladribine and its combination therapy are effective in patients with relapsed and refractory AML and de novo AML. The NCCN guidelines recommend the combination of cladribine as a category 1 recommendation for newly-diagnosed and refractory or relapsed adult AML. Several studies have confirmed the use of Cladribine in the treatment of refractory and relapsed AML.

The strong synergistic anti-cancer effect of HDACi combined with Cladribine has been shown in many cancers such as B-cell chronic lymphocytic leukemia, colon cancer, multiple myeloma, natural killer large granular lymphocytic leukemia, B-cell non-Hodgkin's lymphoma, and mantle cell lymphoma. Our previous study found a synergistic effect on combination of Chidamide and Cladribine in AML cell lines and primary cells. In clinical observation, refractory and relapsed AML patients also responded well to the combination of Chidamide plus Cladribine regimen. This provides a theoretical and practical basis for the use of the combination of Chidamide and Cladribine in AML patients.

DETAILED DESCRIPTION:
This study is aimed to observe the efficacy and safety of the Chidamide Plus Cladribine regimen in treating patients with refractory or relapsed AML. Patients must provide written informed consent and meet all the inclusion criteria and none of the exclusion criteria to be eligible. The eligible patients with refractory or relapsed AML will receive chidamide plus cladribine regimen. Response criteria will be assessed according to the guidelines of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in AML. In case of partial remission, the second identical course will be started. In case of complete remission, allogeneic hematopoietic stem cell transplantation will be performed if available. Patients without complete remission after two courses of treatment will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old and less than 75 years old;
* Clinical diagnosis of Relapsed/Refractory AML (non-APL);
* ECOG performance status score 0-3;
* Participant has the ability to understand and willingness to sign a written consent document.

Exclusion Criteria:

* Pregnancy or nursing
* Uncontrolled significant cardiac disorder
* Psychiatric disorder may interfere with his / her compliance with the study protocol
* Known history of intolerance or allergy to any component of the research regimen
* Any condition not suitable for the trial as judged by the study investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Complete Remission (CR) rate | Bone marrow examination will be performed at the end of Cycle 1 (each cycle is 28 days)
  Less than 5 percent of blast cells in bone marrow aspiration is defined as CR.

SECONDARY OUTCOMES:
Incidences of Adverse Events (AEs) | All AEs reported from the time of study drug administration until 30 days after discontinuation of study drug administration will be collected.
  Safety and Tolerability
Overall Survival (OS) | OS is defined as the number of days from the date of the study enrollment to the date of death of any cause with a minimal 12 months of follow up. Subjects that have not died will be censored at the last known date to be alive.
  The overall survival evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Ge, M.D, Ph.D, Study Director — Medicine School of South East University, China
Locations (1):
- Department of Hematology, Zhongda Hospital Southeast University, Institute of Hematology Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No